CLINICAL TRIAL: NCT06111040
Title: Deconstructing Food Parenting Approaches to Obesity Prevention for the Highly Food Motivated Child
Brief Title: Nurturing Needs Study: Parenting Food Motivated Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Baylor College of Medicine (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R01DK132642 (NIH); 30291 (Other: Temple Institutional Review Board)
Record Dates: First submitted 2023-10-26; First posted 2023-11-01 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Parenting; Eating Behavior; Diet, Healthy; Pediatric Obesity
MeSH Terms: conditions — Feeding Behavior; Pediatric Obesity | interventions — Weights and Measures; Eating

STUDY DESIGN:
Intervention Model Description: Family-based, prospective observational study with interventions at the measurement level
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Caregiver-child dyads (Other): A cohort of 205 caregivers and 205 children aged 4-5 years at baseline will be recruited and followed longitudinally for 18 months.
  Interventions: Other: Measurement

INTERVENTIONS:
Other: Measurement — The only interventions are at the measurement level and consist of two behavioral protocols designed to assess children's eating behavior, where food stimuli are provided and children's behavioral responses are recorded.
  Other Names: Eating in the absence of hunger; Relative reinforcing value of food

SUMMARY:
High food motivation among children is trait-like and increases risks of unhealthy dietary intake and obesity. Scientific knowledge of how parenting can best support healthy eating habits and growth among children who are predisposed to overeating is surprisingly limited. This investigation will identify supportive food parenting approaches for obesity prevention that address the needs of highly food motivated children.

DETAILED DESCRIPTION:
High levels of food motivation among young children are heritable, track over time, and associated with elevated risks of unhealthy eating and obesity. Despite significant growth of family-based obesity prevention efforts, the evidence base is remarkably scant on parenting highly food motivated children to prevent obesity and poor dietary outcomes. The goal of this investigation is to generate a robust basic science evidence for parenting highly food motivated children to prevent excessive dietary intakes and body mass index (BMI) gains during the preschool years. Using a prospective cohort design, this investigation follow 205 caregiver/child dyads over 18 months as children transition from preschool to elementary school, when significant numbers of children begin to experience problems of poor diet quality and obesity. Children with varying food motivation will be recruited to understand whether highly food motivated children have different needs than other children. A multi-method approach will use state-of-the-art measures, including ecological momentary assessment, to comprehensively investigate the amount, types, and consistency of food parenting practices (i.e., specific, goal-oriented behaviors) needed to prevent food motivated behaviors, excessive dietary intake, and BMI gains in children. Specifically, the role of structure (i.e., theoretically supportive) and its differentiation from more coercive types of food parenting control will be comprehensively characterized.

ELIGIBILITY:
Inclusion Criteria:

1. Child ages 4 or 5 years at baseline;
2. Parent/ primary caregiver with legal representation (having 50% or more custody of child);
3. Parent/primary caregiver reporting primary responsibility for child feeding outside of childcare (being with child when they are eating at least two times daily);
4. Caregiver with a cell phone that can be used to send and receive text messages. If there is more than one age-eligible child in the family, we will ask the caregiver to pick the index child.

Exclusion Criteria:

1. Parent/primary caregiver <18 years of age;
2. Child history of major food allergies (e.g., peanuts);
3. Child medication use (e.g., insulin), developmental disability (e.g., autism) or medical condition(s) (e.g., diabetes) known to affect food intake and growth;
4. Foster child.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 416 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Excessive dietary intakes | Baseline, 18 months
  Indicators: SFAS intakes and meal/snack sizes estimated from 24-hour dietary recalls
BMI change | Baseline, 18 months
  % of the 50th percentile per age- and sex-specific CDC reference values for BMI on a log scale

SECONDARY OUTCOMES:
Observed food motivated behaviors | Baseline, 18 months
  Indicators: Eating in the absence of hunger and relative reinforcing value of food

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer O Fisher, PhD, Principal Investigator — Temple University; Sheryl O Hughes, PhD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Temple University - Center for Obesity Research and Education, Philadelphia, Pennsylvania
  - USDA/ARS Children's Nutrition Research Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Research data generated by the project will be supported by TUScholarShare (https://scholarshare.temple.edu/), the institutional repository for Temple University. This is a repository service that is managed by the Temple University Libraries and uses Open Repository, an enhanced DSpace platform that is hosted by Atmire. TUScholarShare has been developed with the intent of helping researchers comply with grant-funding agency requirements. It enables dissemination and long-term preservation and curation (management, use, and re-use) of data.
Time Frame: Within two years of completion of the study
Access Criteria: Researchers will work with the University Libraries Research Data Management Services staff to facilitate the deposit of data into TUScholarShare, and to ensure appropriate metadata and complete documentation of the data to maximize the ability to understand and reuse the data. The data will be published in TUScholarShare for long-term preservation, using services such as file format migration where possible, persistent identifiers (DOIs), persistent Web addresses (handles), and checksums.
  TUScholarShare data resides in two locations, a local Isilon storage system and an off-site cloud-based service, Open Repository. Open Repository's AWS cloud storage service provides extended infrastructure, which includes a production server, test server, fallback servers, data backups, and full system backups
URL: https://scholarshare.temple.edu/

REFERENCES:
- [Background] Buttner C, Skupin A, Reimann T, Rieber EP, Unteregger G, Geyer P, Frank KH. Local production of interleukin-4 during radiation-induced pneumonitis and pulmonary fibrosis in rats: macrophages as a prominent source of interleukin-4. Am J Respir Cell Mol Biol. 1997 Sep;17(3):315-25. doi: 10.1165/ajrcmb.17.3.2279. PMID 9308918